CLINICAL TRIAL: NCT03783143
Title: Serosurvey for Prevalence and Incidence of Lassa Virus Infection in Southern Mali
Brief Title: Prevalence and Incidence of Lassa Virus Infection in Southern Mali
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999919029; 19-I-N029
Record Dates: First submitted 2018-12-19; First posted 2018-12-20 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07-17

CONDITIONS: Lassa Virus Infection
Keywords: Febrile; Human; Lassa Fever; Seroconversion; Natural History
MeSH Terms: conditions — Lassa Fever; Fever; HIV Seropositivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Clinical Cohort: This study population will consist of patient volunteers that visit one of our clinical sites with an undiagnosed febrile illness.
- Cross-sectional Cohort: This study population will consist of patient volunteers that visit one of our clinical sites with an undiagnosed febrile illness.

SUMMARY:
Background:

The disease Lassa fever mostly affects people in Western Africa. It is very similar to other diseases that cause fever, like malaria and yellow fever. People get Lassa fever from mice infected with Lassa virus. It can also be spread from body fluids of people with the disease. Researchers want to learn more about this virus in Mali so they can develop better tools to diagnose and prevent it.

Objective:

To find out how many people in certain areas of southern Mali have ever had Lassa fever and count how many people get the disease every year.

Eligibility:

People ages 6 months to 99 years who live in certain areas of Mali

Design:

Women who are could become pregnant will have a urine pregnancy test at each visit.

Participants will be asked questions about their age, if they have ever had a fever, and if they have ever seen mice in or around their home. This will take about 20 minutes.

Participants will give a blood sample using a needle in a vein in the arm. Young children will give it by pricking a finger or heel with a needle.

Patients with a fever illness will have a medical history and physical exam. They will give blood and nasal swabs 3 times over 21 days.

Participants may be asked to come back 1 time each year for up to 3 more years to take another sample of blood and answer more questions.

DETAILED DESCRIPTION:
In West Africa, as many as 300,000 people are infected annually with Lassa virus (LASV), resulting in approximately 5,000 deaths. Most commonly, human infection comes from contact with infected rodent hosts (Mastomys natalensis), or ingestion or inhalation of virus-laden particles. Person-to-person transmission is also well documented and can cause outbreaks, especially in nosocomial settings. Infection in pregnancy, especially the third trimester, is particularly severe, with maternal mortality rates estimated at 20% and fetal mortality rates nearing 100%. A survey of rodents captured in the village of Soromba (rural commune of Sibirila, district of Bougouni, Mali) found that 25% of M. natalensis had evidence of LASV infection. A 2015 study of LASV infection in the human populations of this region showed seroprevalence of 33.2% and annual incidence rate of 6.3% in 2016.

The purpose of this serosurvey study is to determine the prevalence and incidence of human exposure to LASV in the administrative districts of Bougouni, Yanfolila, and Kolondieba in southern Mali. The study involves 2 separate sub-studies. Study 1 is a cross-sectional serosurvey of residents of the general population selected from a census. The study will follow up to 500 participants at each of 4 study sites (Fakola, Bamba, Filamana, and Guelelinkoro). Participants will be asked to give blood samples at baseline and annually for up to 3 years. Study 2 is a clinic-based serosurvey conducted at local health centers following up to 500 participants per year at each of the 4 study sites (Fakola, Bamba, Filamana, and Guelelinkoro). Patients who report with febrile illness suggestive of Lassa fever will be asked to give blood and nasal swab samples, then return for follow-up visits 5 and 21 days later for clinical consultation and additional blood and swab collection.

All participants will be provided with free medical treatment according to local standard of care as needed for the duration of the study. They will be followed passively between study visits and instructed to report to their local health center if they have a fever. Study visits will be conducted through a common end date, up to 3 years.

Blood and nasal swab samples will be used to identify history of or current LASV infection and for exploratory studies into the biochemistry and pathophysiology of LASV infection. Elucidating the prevalence of LASV infection in the populations of southern Mali may help Malian authorities improve surveillance, and additional research may help develop diagnostics and treatment.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age greater than or equal to 6 months to 99 years.
  2. Resident of one of the study sites for at least 3 months.
  3. Able to provide informed consent.
  4. Agrees to allow storage of samples for future research.

Additional inclusion criteria for the cross-sectional study (study 1):

1. No plans to relocate before the study end date.

Additional inclusion criteria for the clinic-based study (study 2):

1. Has fever (temperature greater than or equal to 38 degree celcius), or has had antecedent of fever for at least 2 consecutive days at the time of screening.
2. One or more of the following:

   1. Excluded typhoid fever and and has at least 1 of the following symptoms: chest pain, sore throat, headache, muscle pain,vomiting, and diarrhea.
   2. Shows bleeding or facial edema.
   3. Does not respond to anti-malarials or antibiotics after 2 days of treatment.
   4. Had contact with a confirmed LF case within the last 3 weeks.

EXCLUSION CRITERIA:

General exclusion criteria:

1. Any condition that, in the opinion of the investigator, contraindicates participation in this study, including conditions that could hinder compliance or that could place participants or study staff at increased risk.
2. Pregnancy.

Additional exclusion criteria for the clinic-based study (study 2):

1. Signs or symptoms of fever-associated conditions other than LF, such as urinary tract infection, or any other infection that may cause fever.

Co-enrollment guidelines: Participants may be co-enrolled in other studies; however, study staff should be notified of co-enrollment

Ages: 6 Months to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals will be randomly identified from village census lists, and a member of the study team will contact the individual by phone or in person about potential participation in the study. In accordance with cultural practices, the individual s entire household will be invited to participate
Sampling Method: Probability Sample
Enrollment: 8524 (Actual)
Dates: Start 2020-12-04 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2024-07-25 (Actual)

PRIMARY OUTCOMES:
Determine the prevalence and | At time of study start
  Determine the prevalence and annual incidence of seroconversion to LASV infection in the general population around each study site in the LASV-endemic area of southern Mali
Determine the incidence of LF in febrile patients attending health centers in southern Mali | Over 3 years
  Determine the incidence of LF in febrile patients attending health centers in southern Mali over 3 years.

SECONDARY OUTCOMES:
Determine the biological, clinical, and virologic parameters of LASV-Soromba infection in study participants with LF. | At time of study start.
  Determine the biological, clinical, and virologic parameters of LASV-Soromba infection in study participants with LF.

CONTACTS AND LOCATIONS:
Overall Officials: Heinrich U Feldmann, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- Icer/Mrtc/Fmos/Usttb, Bamako, Mali

IPD SHARING:
Plan to Share IPD: No
Although samples were collected prospectively all testing is performed retrospectively. Our agreement with the local health centers is to inform them of the overall results of the study and their region in particular. We do not plan to inform individuals.